CLINICAL TRIAL: NCT01225107
Title: A Randomized, Double-Blind, Placebo-Controlled Study of the Effect of Cranberry Extract on the Incidence of Infections in Burn Patients
Brief Title: Effect of Cranberry Extract on Infections in Burn Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Elizabeth Regional Medical Center (Other)
Responsible Party: David Voigt, Saint Elizabeth Regional Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 609-052
Record Dates: First submitted 2010-08-11; First posted 2010-10-20 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Burn
Keywords: Burns; Infections; Cranberry
MeSH Terms: conditions — Burns; Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inert Placebo Capsule (Placebo Comparator)
  Interventions: Drug: Inert Placebo Capsule
- Cranberry Extract (Experimental)
  Interventions: Dietary Supplement: Cranberry Extract

INTERVENTIONS:
Dietary Supplement: Cranberry Extract — 500mg TID
  Other Names: Cranberry
  Arms: Cranberry Extract
Drug: Inert Placebo Capsule — Inert substance, 3 times per day in capsule form
  Arms: Inert Placebo Capsule

SUMMARY:
Bacterial infections are a common complication in patients suffering from burns. These infections can cause significant morbidity and often mortality. Antimicrobial resistance coupled with the prevalence of burn-related infections warrants the identification of alternative substances in the treatment of burn-related infections. The cranberry has been examined as a potential agent in the prevention of other types of infections and it appears to have anti-adherence effects on bacteria. In addition, the cranberry has demonstrated general inhibitory effects against some types of bacteria suggesting that it may be a useful agent in the prevention of bacterial infections in burn patients. The purpose of the present study is to investigate the effect of cranberry extract on the incidence of infections in burn patients.

DETAILED DESCRIPTION:
Methods

Design. The present study is a prospective, randomized, double-blind, placebo-controlled study of the effect of taking three times daily doses of cranberry extract in capsule form on the incidence of infection in burn patients.

Participants. Eighty patients suffering from burns and admitted to the Saint Elizabeth Regional Medical Center Burn Center, Lincoln, NE will take place in the proposed study.

Inclusion Criteria. Patients will be asked to participate in the study if the following criteria are met:

* Patients are admitted to the Saint Elizabeth Regional Medical Center Burn Unit.
* Age 19 and older.
* Patients have an expected hospital stay of 7 days or more.
* Patients are able to consume oral medication capsules.

Exclusion Criteria. Patients will not be asked to participate in the study if any of the following are present:

* Patients have a known infection.
* Patients are not able to consume oral medication capsules.
* Patients have any known allergies to cranberry or placebo components.
* Patients have known allergy to aspirin (cranberries may contain salicylic acid).
* Patients are pregnant or breast-feeding.
* Patients are taking warfarin
* Patients with known nephrolithiasis.
* Patients with renal impairment as evidenced by a creatinine clearance that is less than predicted by Cockroft-Gault formula.

A cranberry extract standardized by Ocean Spray Cranberries, Inc. will be placed into capsules in the Saint Elizabeth Regional Medical Center pharmacy. Each cranberry capsule will contain 500mg of cranberry extract. Placebo capsules will be made to look identical to cranberry capsules and will also be made at the Saint Elizabeth Regional Medical Center pharmacy. A staff pharmacist will separate the capsules into a cranberry extract group and a placebo group. A staff pharmacist will randomly assign patients to either the cranberry extract group or the placebo group. The patient, physicians, and research staff involved in data collection will be blinded to patient group assignment.

Procedure. After admission to the burn unit and after the physician has deemed that the patient is able to consume medication capsules orally, patients meeting all other selection criteria will be asked to participate in the study. Study rationale and procedures will be described to patients and informed consent will be obtained if patients indicate a willingness to participate. Basic demographic data, burn/wound related information and information pertaining to any other infections will be obtained. Participants will be randomly assigned to either the placebo or the cranberry group. Participants will be given one capsule as soon as possible after hospital admission (or as soon as they have been deemed capable of consuming medication capsules orally) and then as close as possible to 8 hours after the first dose. Patients will then be placed on an 8 hour dosing schedule (i.e., one capsule every 8 hours). Burn wounds will be examined for any clinical signs of infection as judged by attending physician on a daily basis. The determination as to whether an infection is present vs. absent will be made by a physician utilizing specific criteria. If signs of infection are present, cultures of the wound site will be taken and bacterial type will be recorded. After initial infection, wound sites will be observed to determine if infections resolve with treatment. If treatment does not seem to eradicate the infection, another bacterial culture will be taken and bacterial analysis will be performed and recorded. Data pertaining to wound infection and wound appearance will be taken on a daily basis throughout the duration of the patient's hospital stay. In addition, information pertaining to all infections present in each patient will be recorded on a daily basis throughout the patient's entire hospital stay. The determination as to whether other infections are present vs. absent will be made by a physician utilizing specific criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patients are admitted to the Saint Elizabeth Regional Medical Center Burn Unit.
* Age 19 and older.
* Patients have an expected hospital stay of 7 days or more.
* Patients are able to consume oral medication capsules.

Exclusion Criteria:

* Patients have a known infection.
* Patients are not able to consume oral medication capsules.
* Patients have any known allergies to cranberry or placebo components.
* Patients have known allergy to aspirin (cranberries may contain salicylic acid).
* Patients are pregnant or breast-feeding.
* Patients are taking warfarin
* Patients with known nephrolithiasis.
* Patients with renal impairment as evidenced by a creatinine clearance that is less than predicted by Cockroft-Gault formula.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Overall Infection Rate | average of 17 days
  Patients will be enrolled in the study throughout the duration of their hospital stay. They will be assessed on a daily basis.

SECONDARY OUTCOMES:
Time between study enrollment and acquisition of infection | average of 17 days
  Patients will be enrolled in the study throughout the duration of their hospital stay. They will be assessed on a daily basis.

CONTACTS AND LOCATIONS:
Overall Officials: David W Voigt, M.D., Principal Investigator — Saint Elizabeth Regional Medical Center
Locations (1):
- Saint Elizabeth Regional Medical Center, Lincoln, Nebraska, United States